CLINICAL TRIAL: NCT04953468
Title: Study on the Mechanism of the Expression of ANXA2 in the Extracellular Space in the Microenvironment of Periumoral Edema to Promote Glioma Invasion
Brief Title: Expression of ANXA2 in the Extracellular Space in the Microenvironment of Periumoral Edema Promotes Glioma Invasion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021020
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Glioma
Keywords: glioma; ANXA2 Expression; periatumoral edema zone
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Immunohistochemistry of glioma tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ANXA2 high expression in glioma: We plan to grade the dyeing intensity of ANXA2 as follows: level 0 for non-stained, level 1 for lighter colored, level 3 for dark brown, and level 2 for those between the latter two.We planned to divide the staining proportion into 5 grades: grade 0 for those without staining, grade 1 for those with staining proportion < 10%, grade 2 for those with staining proportion ≥10% and < 50%, grade 3 for those with staining proportion ≥50% and < 80%, and grade 4 for those with staining proportion ≥ 80%.Finally, staining intensity grading × staining proportion grading = expression level was calculated In glioma tissues, samples with expression level ≥6 points were identified as the ANXA2 high expression group
  Interventions: Diagnostic Test: expression level of ANXA2 protein
- ANXA2 low expression in glioma: We plan to grade the dyeing intensity of ANXA2 as follows: level 0 for non-stained, level 1 for lighter colored, level 3 for dark brown, and level 2 for those between the latter two.We planned to divide the staining proportion into 5 grades: grade 0 for those without staining, grade 1 for those with staining proportion < 10%, grade 2 for those with staining proportion ≥10% and < 50%, grade 3 for those with staining proportion ≥50% and < 80%, and grade 4 for those with staining proportion ≥ 80%.Finally, staining intensity grading × staining proportion grading = expression level was calculated In glioma tissues, samples with expression level <6 points were identified as the ANXA2 low expression group
  Interventions: Diagnostic Test: expression level of ANXA2 protein
- ANXA2 high expression in PTBE: We plan to grade the dyeing intensity of ANXA2 as follows: level 0 for non-stained, level 1 for lighter colored, level 3 for dark brown, and level 2 for those between the latter two.We planned to divide the staining proportion into 5 grades: grade 0 for those without staining, grade 1 for those with staining proportion < 10%, grade 2 for those with staining proportion ≥10% and < 50%, grade 3 for those with staining proportion ≥50% and < 80%, and grade 4 for those with staining proportion ≥ 80%.Finally, staining intensity grading × staining proportion grading = expression level was calculated In PTBE, samples with expression level ≥2 were regarded as the ANXA2 high expression group
  Interventions: Diagnostic Test: expression level of ANXA2 protein
- ANXA2 low expression in PTBE: We plan to grade the dyeing intensity of ANXA2 as follows: level 0 for non-stained, level 1 for lighter colored, level 3 for dark brown, and level 2 for those between the latter two.We planned to divide the staining proportion into 5 grades: grade 0 for those without staining, grade 1 for those with staining proportion < 10%, grade 2 for those with staining proportion ≥10% and < 50%, grade 3 for those with staining proportion ≥50% and < 80%, and grade 4 for those with staining proportion ≥ 80%.Finally, staining intensity grading × staining proportion grading = expression level was calculated In PTBE, samples with expression level <2 were regarded as the ANXA2 low expression group
  Interventions: Diagnostic Test: expression level of ANXA2 protein

INTERVENTIONS:
Diagnostic Test: expression level of ANXA2 protein — The expression level of ANXA2 protein in glioma and PTBE was detected by immunohistochemistry

SUMMARY:
The prognostic value of ANXA2 expression in tumor tissue and PTBE was analyzed, so as to seek new therapies to inhibit glioma invasion and improve the prognosis of glioma patients

DETAILED DESCRIPTION:
The main reason for the poor prognosis of glioma is the invasion of tumor cells along the extracellular space (ECS) in the periatumoral edema zone (PTBE).Previous studies have shown that ANXA2 is highly expressed in glioma and promotes tumor growth and invasion, while its expression in the PTBE microenvironment of glioma and its mechanism of action on tumor invasion have not been reported.Previous study found that ANXA2 was overexpressed in gliomas and was associated with poor prognosis, and the low expression of ANXA2 significantly inhibited tumor invasion in vitro.Relevant studies have also confirmed that as an exocrine protein, it mainly plays a role in ECS, and it has previously been carried out on the tissue structure of ECS in tumor microenvironment.Therefore, investigators planned to study the mechanism of ANXA2 expression in PTBE microenvironment ECS on tumor invasion.This project aims to take glioma related issues as the research object and analyze tumor tissue and tumor tissue

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone microneurosurgical resection of the tumor in our hospital and are pathologically confirmed to be supratentorial glioma;
* Preserving the remaining tissue samples of paired gliomas and PTBE for pathological examination;
* The patients agreed to be enrolled and signed the informed consent;
* The clinical data of the patients are complete and not lost;
* No serious complications occurred after surgery.

Exclusion Criteria:

* All glioma patients who did not meet the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18-75 years) who underwent microsurgical resection of glioma in the Neurosurgery Department of Peking University Third Hospital between 2018 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of surgery to the date of death from any cause, assessed up to 18 weeks.
  Follow-up information was collected by telephone follow-up and regular review when patients returned to the hospital. Telephone follow-up was conducted every 3 months, and the main follow-up content was survival time, and the end point of follow-up was to the patient's death

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jun, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No